CLINICAL TRIAL: NCT04394429
Title: Analysis of Events of Endotracheal Tube Obstruction in Covid-19 Patients Requiring Mechanical Ventilation
Brief Title: Endotracheal Tube Obstruction in Covid-19 Patients Requiring Mechanical Ventilation
Acronym: TubeObs-Covid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7803
Record Dates: First submitted 2020-05-18; First posted 2020-05-19 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-05

CONDITIONS: Sars-CoV2
Keywords: Endotracheal Tube; ETT; Intubation; Mechanical ventilation; Endotracheal tube obstruction; ICU; Covid-19; SARS-CoV-2; ARDS
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The COVID-19 pandemic is very present in our region, the Grand-Est region is considered as one of the first COVID-19 epicentres in France. COVID-19 causes an acute respiratory distress syndrome requiring prolonged mechanical ventilation in resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Major Subject (≥18 years)
* Subject with COVID 19 (radiological suspicion or microbiological confirmation)
* Subject hospitalised in the intensive care unit at the NHC of the University Hospitals of Strasbourg between 01/03/2020 and 03/04/2020.
* Subject treated by mechanical ventilation
* Subject who has not expressed his opposition, after information, to the re-use of his data for the purposes of this research

Translated with www.DeepL.com/Translator (free version)

Exclusion Criteria:

* Subject who expressed opposition to participating in the study
* Subject under guardianship, curatorship or safeguarding of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subject with COVID 19 hospitalized in the intensive care unit at the NHC of the University Hospitals of Strasbourg
Sampling Method: Non-Probability Sample
Enrollment: 184 (Estimated)
Dates: Start 2020-04-24 (Actual); Primary Completion 2021-06-24 (Estimated); Study Completion 2021-06-24 (Estimated)

PRIMARY OUTCOMES:
Analysis of risk factors for intubation tube obstruction | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Bob HEGER, Study Director — Anesthesia-Resuscitation Department - Strasbourg University Hospitals
Locations (1):
- Service d'Anesthésie-Réanimation - Nouvel Hôpital Civil, Strasbourg, France